CLINICAL TRIAL: NCT00975221
Title: A Randomized Double-blind Placebo-controlled Study to Evaluate the Efficacy and Safety of Cinacalcet for the Treatment of Hypercalcemia in Subjects With Primary Hyperparathyroidism Unable to Undergo Parathyroidectomy
Brief Title: Efficacy and Safety Study of Cinacalcet for the Treatment of Hypercalcemia in Patients With Primary Hyperparathyroidism Unable to Undergo Parathyroidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070277
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Hyperparathyroidism, Primary; Hypercalcemia
Keywords: Primary hyperparathyroidism; Parathyroidectomy; Hypercalcemia
MeSH Terms: conditions — Hyperparathyroidism, Primary; Hypercalcemia | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinacalcet (Experimental): Participants received cinacalcet at a starting dose of 30 mg orally BID and were eligible for a dose titration once every 3 weeks during the 12-week dose-titration phase based on corrected total serum calcium concentration and safety assessments. Participants continued to receive cinacalcet for another 16 weeks during the efficacy assessment phase and then continued into the open-label extension phase and received cinacalcet at a starting dose of 30 mg BID for 24 weeks. The dose of cinacalcet could have been increased or decreased as needed to maintain a corrected total serum calcium concentration within the normal range through Week 52.
  Interventions: Drug: Cinacalcet
- Placebo (Placebo Comparator): Participants received placebo orally twice a day (BID) for 12 weeks during the dose titration phase and for another 16 weeks during the efficacy assessment phase. Participants then continued into the open-label extension phase and received cinacalcet at a starting dose of 30 mg BID for 24 weeks. The dose of cinacalcet could have been increased or decreased as needed to maintain a corrected total serum calcium concentration within the normal range through Week 52.
  Interventions: Drug: Cinacalcet; Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — Administered orally at a starting dose of 30 mg twice a day (BID). Participants will be eligible for a dose titration once every 3 weeks during the placebo-controlled dose titration phase based on corrected total serum calcium concentration and safety assessments obtained the previous week. Doses may be sequentially increased to 60 mg BID, 90 mg BID, and 90 mg 3 times a day (TID).
  Other Names: Sensipar; Mimpara
Drug: Placebo — Administered orally following the same tiitration regimen as the experimental arm.
  Arms: Placebo

SUMMARY:
This study is designed to demonstrate the efficacy and to assess the safety of cinacalcet for the reduction of hypercalcemia in patients with primary hyperparathyroidism for whom parathyroidectomy is indicated on the basis of an elevated corrected total serum calcium, but who are unable to undergo parathyroidectomy.

DETAILED DESCRIPTION:
The study will consist of a 30-day screening phase, a 12-week placebo-controlled dose-titration phase, and a 16-week placebo-controlled efficacy assessment phase (EAP). Participants who complete 28 weeks on study will continue into an open-label safety extension phase for 24 weeks of investigational cinacalcet treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of primary hyperparathyroidism (HPT)
* subjects must have the following laboratory values:

  1. local/historical laboratory result showing a corrected total serum calcium > 1 mg/dL (0.25 mmol/L) above the upper limit of normal and

     ≤ 12.5 mg/dL (3.12 mmol/L) within the past 12 months, and
     * local/historical laboratory result showing a plasma parathyroid horone (PTH) > 75% of upper limit of normal within the past 12 months, and
     * one central laboratory draw at the screen visit showing a corrected total serum calcium > 11.3 mg/dL (2.82 mmol/L) and ≤ 12.5 mg/dL (3.12 mmol/L), and
     * one central laboratory draw at the screen visit showing a plasma PTH > 55 pg/mL (5.8 pmol/L) OR
  2. two central laboratory draws performed during the screening period at least 7 days apart, showing a

     * corrected total serum calcium > 11.3 mg/dL (2.82 mmol/L) and ≤ 12.5 mg/dL (3.12 mmol/L), and
     * plasma PTH > 55 pg/mL (5.8 pmol/L)
* not able to undergo parathyroidectomy for ≥ 1 of the following reasons:

  * failed parathyroidectomy
  * comorbid conditions contraindicating parathyroidectomy
  * parathyroidectomy not considered appropriate or is not feasible by primary physician and subject
* before any study-specific procedure is performed, the appropriate written informed consent must be obtained

Exclusion Criteria:

* symptoms attributable to hypercalcemia, requiring immediate medical intervention, as judged by the investigator (including acute kidney stone, nausea and vomiting requiring intravenous hydration, confusion, lethargy, stupor, or coma)
* unstable medical condition, defined as having been hospitalized within 30 days before the date of informed consent, or otherwise unstable in the judgment of the investigator
* administration of drugs that increase serum calcium concentration, including but not limited to thiazide diuretics or lithium
* initiated bisphosphonate therapy or changed bisphosphonate dose within 12 weeks before the date of informed consent
* current administration of drugs for ventricular arrhythmia
* unable to provide informed consent, or is at risk for poor compliance with study procedures
* currently enrolled in another investigational device or drug study(s), or completed such study within 30 days before the date of informed consent
* known hypersensitivity to or unable to tolerate cinacalcet
* received treatment with cinacalcet within 60 days before the date of informed consent
* history of seizures or an adjustment of anti-seizure medication within 12 weeks before the date of informed consent
* family history or diagnosis a genetic syndrome, such as familial benign hypocalciuric hypercalcemia (FBHH) or multiple endocrine neoplasia type 1 (MEN1) and type 2 (MEN2), where primary HPT is one of the clinical manifestations of familial benign hypocalciuric hypercalcemia (FBHH)
* refused to use highly effective contraceptive measures (as determined by the investigator) throughout the study
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-03-10 (Actual); Primary Completion 2012-07-12 (Actual); Study Completion 2012-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (22):
  - Research Site, Lake Forest, California
  - Research Site, Lancaster, California
  - Research Site, Los Gatos, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Weston, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Kenner, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Morehead City, North Carolina
  - Research Site, Columbus, Ohio
- Australia (5):
  - Research Site, Randwick, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Footscray, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Nedlands, Western Australia
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, London, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Toronto, Ontario
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Szeged
- Research Site, Warsaw, Poland
- Portugal (2):
  - Research Site, Coimbra
  - Research Site, Lisbon
- Russia (4):
  - Research Site, Moscow
  - Research Site, Rostov-na-Dony
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl

REFERENCES:
- [Background] Khan A, Bilezikian J, Bone H, Gurevich A, Lakatos P, Misiorowski W, Rozhinskaya L, Trotman ML, Toth M. Cinacalcet normalizes serum calcium in a double-blind randomized, placebo-controlled study in patients with primary hyperparathyroidism with contraindications to surgery. Eur J Endocrinol. 2015 May;172(5):527-35. doi: 10.1530/EJE-14-0877. Epub 2015 Jan 30. PMID 25637076
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 29 centers in United States, Australia, Canada, Hungary, Poland, Portugal, and Russian Federation.
  The first participant enrolled on 10 March 2010 and the last participant enrolled on 28 December 2011.
Pre-assignment Details: This study consisted of a 12-week placebo-controlled dose-titration phase, a 16-week placebo-controlled efficacy assessment phase (EAP), and an open-label safety extension phase for 24 weeks of cinacalcet treatment. Participants were randomized in a 1:1 ratio to cinacalcet or placebo stratified by bisphosphonate use.
Period: Titration Phase (Weeks 1-12)
Arm/Group | Placebo | Cinacalcet
Started | 34 | 33
Received Study Drug | 34 | 33
Completed | 31 | 29
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Requirement for alternative therapy | 1 | 0
Not completed — Other | 0 | 1
Period: Efficacy Assessment Phase (Weeks 13-28)
Arm/Group | Placebo | Cinacalcet
Started | 30 (1 participant who completed the Titration Phase did not enter the EAP) | 29
Completed | 30 | 28
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Open-label Extension Phase (Weeks 29-52)
Arm/Group | Placebo | Cinacalcet
Started | 29 (1 participant who completed the EAP did not enter the open-label phase) | 28
Completed | 27 | 27
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cinacalcet | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (8.9) | 69.5 (13.0) | 72.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 4 | 5
  Hispanic or Latino | 0 | 1 | 1
  White or Caucasian | 33 | 28 | 61
Albumin-corrected Calcium [Mean (Standard Deviation); unit: mg/dL] | 11.80 (0.48) | 11.73 (0.45) | 11.77 (0.46)
Intact Parathyroid Hormone (iPTH) [Mean (Standard Deviation); unit: pg/mL] | 238.6 (212.2) | 179.0 (98.0) | 209.7 (168.4)
Bisphosphonate Use [Number; unit: participants]
  Yes | 10 | 9 | 19
  No | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Mean Corrected Total Serum Calcium Concentration ≤ 10.3 mg/dL (2.57 mmol/L) During the EAP
Time Frame: Efficacy assessment phase (study visits at Weeks 16, 20, 24, and 28)
Population: Full analysis set (all participants randomized to treatment). For participants with no data for the EAP, the last post-baseline value from the titration phase was used to impute the missing EAP values (last value carried forward (LVCF) imputation). Participants with only baseline information were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 34 | 33
percentage of participants | 0.0 | 75.8
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) statistic = 39.866

2. Secondary Outcome: Percentage of Participants With a ≥ 1 mg/dL (0.25 mmol/L) Decrease From Baseline in Mean Corrected Total Serum Calcium Concentration During the EAP
Time Frame: Baseline and the EAP (mean of Weeks 16, 20, 24, and 28)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 34 | 33
percentage of participants | 5.9 | 84.8
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH statistic = 40.953

3. Secondary Outcome: Percent Change From Baseline in Corrected Total Serum Calcium Concentration During the EAP
Time Frame: Baseline and the EAP (mean of Weeks 16, 20, 24, and 28)
Population: Full analysis set with at least 1 post-baseline measurement; for participants with no data for the EAP, the last post-baseline value from the titration phase was used to impute the missing EAP values (LVCF imputation).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 33 | 33
percent change | -1.66 (0.99) | -15.21 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) with baseline corrected serum calcium and baseline bisphosphonate included as covariates; LS Mean Treatment Difference = -13.55, 95% CI 2-sided [-16.23 to -10.88], Standard Error of Mean 1.34 — Treatment difference: cinacalcet-placebo

4. Secondary Outcome: Percent Change From Baseline in Plasma Parathyroid Hormone Level During the EAP
Time Frame: Baseline and the EAP (mean of Weeks 16, 20, 24, and 28)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Cinacalcet
Number analyzed (Participants) | 33 | 31
percent change | -1.01 (4.05) | -23.80 (4.18)
Statistical Analysis 1: Comparison: Placebo vs Cinacalcet; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Treatment Difference = -22.79, 95% CI 2-sided [-34.01 to -11.57], Standard Error of Mean 5.61 — Treatment difference: cinacalcet-placebo

ADVERSE EVENTS:
Time Frame: 60 Weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Double-blind Phase: Placebo: Participants received placebo orally twice a day (BID) for 12 weeks during the dose titration phase and for another 16 weeks during the efficacy assessment phase.
- Double-blind Phase: Cinacalcet: Participants received cinacalcet at a starting dose of 30 mg orally BID and were eligible for a dose titration once every 3 weeks during the 12-week double-blind dose-titration phase based on corrected total serum calcium concentration and safety assessments. Participants continued to receive cinacalcet for another 16 weeks during the double-blind efficacy assessment phase.
- Open-label Phase: Previous Placebo: Participants who received placebo during the double-blind phase (Weeks 1-28) then received cinacalcet at a starting dose of 30 mg BID for 24 weeks in the open-label extension phase. The dose of cinacalcet could have been increased or decreased as needed to maintain a corrected total serum calcium concentration within the normal range through Week 52.
- Open-label Phase: Previous Cinacalcet: Participants who received cinacalcet during the double-blind phase continued to receive cinacalcet at a starting dose of 30 mg BID for 24 weeks in the open-label extension phase. The dose of cinacalcet could have been increased or decreased as needed to maintain a corrected total serum calcium concentration within the normal range through Week 52.
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Cinacalcet | Open-label Phase: Previous Placebo | Open-label Phase: Previous Cinacalcet
Serious Adverse Events (participants affected / at risk) | 4/34 | 3/33 | 7/29 | 1/28
Other Adverse Events (participants affected / at risk) | 15/34 | 25/33 | 15/29 | 10/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Placebo (N=34) | Double-blind Phase: Cinacalcet (N=33) | Open-label Phase: Previous Placebo (N=29) | Open-label Phase: Previous Cinacalcet (N=28)
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Placebo (N=34) | Double-blind Phase: Cinacalcet (N=33) | Open-label Phase: Previous Placebo (N=29) | Open-label Phase: Previous Cinacalcet (N=28)
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 6 | 9 | 6 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 2 | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 6 | 4 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 2
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.